CLINICAL TRIAL: NCT04207086
Title: A Phase II, Open Label, Single Arm Study of Neoadjuvant Pembrolizumab and Lenvatinib for Patients With Resectable Stage III Melanoma
Brief Title: A Phase II Study of Neoadjuvant Pembrolizumab & Lenvatinib for Resectable Stage III Melanoma
Acronym: Neo PeLe
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIA/CT2019/281; OTSP 57111 (Other: Merck Sharp & Dohme)
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Melanoma Stage III
Keywords: Neoadjuvant therapy; Adjuvant therapy; Pembrolizumab; Lenvatinib; Pathological response; RECIST response; Metabolic response; Translational research
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 wk pembrolizumab & lenvatinib, surgery, 46 wk pembrolizumab (Experimental): Neoadjuvant pembrolizumab & lenvatinib for 6 weeks followed by definitive surgery then adjuvant pembrolizumab alone for 46 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda
Drug: Lenvatinib — Lenvatinib is an oral potent multiple RTK inhibitor that selectively inhibits VEGF receptors, VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4), fibroblast growth factor receptor (FGFR1-4), platelet derived growth factor (PDGFRα), stem cell factor receptor (KIT), and rearranged during transfection (RET).
  Other Names: Lenvima

SUMMARY:
In many cancers, early stage diagnosis and early treatment offers the best chance of a prolonged recurrence free- and overall survival. In stage III/IV resectable melanoma, an opportunity exists to improve outcomes with the addition of neoadjuvant and adjuvant systemic therapy as an adjunct to surgery. Neoadjuvant clinical trials for resectable but bulky stage III/IV melanoma allows for the efficient and rapid evaluation of drug activity in humans utilising multiple clinical endpoints of metabolic, radiological and pathological response; relapse-free survival; overall survival.

DETAILED DESCRIPTION:
New therapeutic strategies for melanoma come as a result of significant advances in the understanding of the immunomodulatory mechanisms and molecular biology. The resulting new therapeutic strategies include oncogene-targeted therapy and immune checkpoint blockade, and these are now approved therapies that have transformed the routine clinical management for patients with metastatic disease. However, most patients with advanced melanoma still die of their disease, and thus, there remains an urgent need to improve upon current therapies. Most patients with advanced disease eventually progress, and the question as to whether earlier treatment with systemic therapy after resection of all macroscopic melanoma (adjuvant therapy) improves long term survival is under investigation in melanoma and other solid malignancies. Furthermore, with the increased number of therapies utilised in melanoma, the question of optimal sequencing and selection of single or combination therapy remains unanswered.

Neoadjuvant clinical trials in patients with resectable but bulky stage III/IV melanoma allows for the rapid evaluation of drug activity in humans utilising multiple clinical endpoints (metabolic response with Positron Emission Tomography [PET], clinical response with Computed Tomography [CT] imaging, pathological response, relapse-free survival and overall survival) and translational endpoints (morphological, genetic and immunophenotyping of tumour and blood).

This trial will test the combination of pembrolizumab and lenvatinib as neoadjuvant and pembrolizumab as adjuvant therapy for twenty adult patients with histologically confirmed RECIST 1.1 measurable and resectable AJCC (8th edition) Stage IIIB, IIIC or IIID cutaneous or unknown primary melanoma.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. Pembrolizumab is a potent humanized immunoglobulin G4 monoclonal antibody with high specificity of binding to the programmed cell death 1 receptor, thus inhibiting its interaction with programmed cell death ligand 1 and programmed cell death ligand 2. Pembrolizumab is indicated for the treatment of patients across a number of indications because of its mechanism of action to bind the PD-1 receptor on the T cell.

Angiogenesis, the formation of new blood vessels from a pre-existing vascular network, is essential for tumour growth and metastasis. Vascular endothelial growth factor (VEGF) and its receptors play a major role in tumour angiogenesis. Lenvatinib is an oral potent multiple RTK inhibitor that selectively inhibits VEGF receptors. In clinical use, lenvatinib is one of the only inhibitors currently labelled with a mechanism of action as an inhibitor of not only VEGFRs but also fibroblast growth factor receptors, both of which are currently believed to very important for tumour angiogenesis. Tumour blood vessels are abnormal, both structurally and functionally, relative to those of non-malignant tissues. Normalizing the tumour vasculature with antiangiogenic agents could potentially be used to improve the effectiveness of immunotherapy, particularly immune checkpoint blockade. The evidence indicates that the potential benefit of such combinations will be manifested though modulation of both the tumour vasculature and the tumour immune microenvironment.

The development of combination therapy of lenvatinib and an anti-PD-1 antibody pembrolizumab is ongoing for various solid tumours. In addition to efficacy and safety endpoints, testing this combination in the neoadjuvant setting provides a valuable opportunity to investigate potential biomarkers and mechanisms of responsiveness, resistance, toxicity and relapse. Limiting the combination of drugs to the neoadjuvant period only, limits the toxicity that may be experienced by patients whilst maintaining an effective treatment regimen.

In many cancers, early stage diagnosis and early treatment offers the best chance of a prolonged recurrence free- and overall survival. In stage III/IV resectable melanoma, an opportunity exists to improve outcomes with the addition of neoadjuvant and adjuvant systemic therapy as an adjunct to surgery. Neoadjuvant clinical trials for resectable but bulky stage III/IV melanoma allows for the efficient and rapid evaluation of drug activity in humans utilising multiple clinical endpoints of metabolic, radiological and pathological response; relapse-free survival; overall survival. Recent clinical trials of neoadjuvant ipilimumab combined with nivolumab (OPACIN-NEO) and neoadjuvant dabrafenib combined with trametinib (NeoCombi) in resectable stage III melanoma showed that a pathological response (< 50% viable tumour at tumour bed in the former trial, and complete response in the latter) was associated with a longer relapse-free survival

The rationale for this study design is therefore based on the hypothesis that six weeks of combined pembrolizumab and lenvatinib may be sufficient to induce an enhanced tumoral immunity to result in a higher pathological and clinical response at the time of definitive surgery.

The clinical and translational findings from this study have the potential to inform rational decisions regarding combinations of treatment both in the metastatic and the adjuvant settings. This is a critical study to inform future practice and future phase 3 clinical trials. The neoadjuvant design provides an important opportunity to address critical translational endpoints from multiple blood draws and tissue biopsies during treatment. From this, the evaluation of potential biomarkers and mechanisms of responsiveness, resistance, toxicity and relapse is possible, beyond the traditional clinical, pathological and radiological parameters. Baseline and serial blood, and tissue samples will be analysed at MIA translational research facilities. The biomarker component of this study will require blood samples and core biopsies of tumour tissue at the following time points:

Baseline (PRE) Week 1 (EDT 1) Week 6 - complete lymph node dissection specimen (POST) At Relapse (RELAPSE) if applicable and available

Neoadjuvant treatment will be administered for 6 weeks, followed by complete resection of tumour to no evidence of disease. Surveillance of disease during the 6 week neoadjuvant period will be undertaken with surgical assessments and with ultrasounds of the affected lymph node basin. Surgery is followed by 46 weeks of pembrolizumab adjuvant therapy or until disease relapse, death, intolerable adverse drug reactions or by withdrawal of patient consent. After 52 weeks of the study treatment phase, patients will be followed 3 monthly for relapse (and progression, following relapse) and survival for 5 years.

The efficacy endpoints for this study have been used across the International Neoadjuvant Melanoma Consortium.

ELIGIBILITY:
Inclusion Criteria:

* 1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* 2. Male/female participants who are at least 18 years of age on the day of signing informed consent.
* 3. Histologically confirmed diagnosis of resectable AJCC (8th edition) Stage IIIB, IIIC or IIID cutaneous or unknown primary melanoma (except for any in-transit or satellite metastases) will be enrolled in this study. Note:

  * At baseline, patients may have a primary melanoma in addition to nodal disease.
  * At baseline, there must be sufficient nodal +/- primary disease which is amenable to multiple excision or core biopsies biopsies.
  * "Resectable" disease is defined as having no significant vascular, central nervous system or bony involvement. Only cases where a complete surgical resection leading to tumour free margins and which is safely achieved is considered "resectable".
* 4. Have measurable disease based on RECIST version 1.1 criteria: ≥ 10mm in the longest diameter for primary (if applicable) lesions and ≥ 15mm in the shortest diameter for lymph nodes.
* 5. Have provided a newly obtained core or excisional biopsy of an affected lymph node lesion which has been not previously irradiated. Archival tissue from the primary melanoma (if applicable) will also be collected, if available, but is not a requirement for study entry.
* 6. Able to swallow and retain oral medication.
* 7. A male participant must agree to use a contraception during the treatment period and for at least and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period and for at least 120 days after the last dose.
* 8. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least and for at least 120 days after the last dose of study treatment.
* 9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of first dose of study treatment.
* 10. Have adequate organ function as defined by routine laboratory testing.
* 11. Adequately controlled blood pressure, with or without anti-hypertensive medications, defined as ≤ 150/90 mmHg at screening and no change in anti-hypertensive medications within one week of the first dose of study treatment. Note: Patients who are taking ≥ 3 anti-hypertensive medications at baseline will require approval from the Lead Investigator prior to enrolment.
* 12. Anticipated life expectancy of > 12 months.

Exclusion Criteria:

* 1. A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to the first dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* 2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
* 3. Has received prior treatment for melanoma including investigational agents within 4 weeks prior to first dose of study treatment. The following are permitted:

  * Surgery for primary or past stage III melanoma.
  * Prior adjuvant interferon or ipilimumab for resected stage II/III melanoma and have recovered to ≤ Grade 1 or baseline from any treatment related adverse effects.
* 4. Has had major surgery within 3 weeks prior to first dose of study treatments. Note: adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility.
* 5. Participants who have not recovered adequately from any toxicity from other anti- cancer treatment regimens.
* 6. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. Prior radiotherapy to the presenting tumour is prohibited.
* 7. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* 8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* 9. Has a diagnosis of immunodeficiency and is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug. The following are permitted:

  * Vitiligo,
  * Type I diabetes mellitus,
  * Residual autoimmune hypothyroidism on stable hormone replacement,
  * Resolved childhood asthma or atopy,
  * Psoriasis not requiring systemic treatment,
  * Autoimmune conditions which are not expected to recur in the absence of an external trigger.
* 10. Has active autoimmune disease that has required systemic treatment in the past 12 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). The following are permitted:

  * Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc, Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if patient on a stable dose,
  * Non-absorbed intra-articular steroid injections are permitted.
* 11. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. The following malignancies, if undergone successful definitive resection or curative treatment, are permitted:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy)
  * Prostatic intraepithelial neoplasia
  * In situ melanoma
  * Atypical melanocytic hyperplasia
  * Multiple primary melanomas
  * Other malignancies for which the patient has been disease free for 1 year.
* 12. Has known CNS metastases and/or carcinomatous meningitis.
* 13. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* 14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis or current interstitial lung disease.
* 15. Has an active infection requiring systemic therapy.
* 16. Has a known history of Human Immunodeficiency Virus (HIV).
* 17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* 18. Has a known history of active TB (Bacillus Tuberculosis).
* 19. Current diagnosis of any gastrointestinal condition that might affect the absorption of lenvatinib (e.g. malabsorption syndrome, gastrointestinal anastomosis, bariatric surgery).
* 20. Has a pre-existing ≥ Grade 3 gastrointestinal or non-gastrointestinal fistula.
* 21. History of, or current cardiovascular disease including: Uncontrolled arrhythmias associated with haemodynamic instability, Uncontrolled arrhythmias requiring medical treatment at screening, Unstable angina within 6 months of the first dose of study drug, myocardial infarction within 6 months of the first dose of study drug

  * >NYHA grade 2 congestive cardiac failure
  * Uncontrolled and treatment refractory hypertension systolic > 150 mmHg and/or diastolic > 90 mmHg in spite of an optimized regimen of antihypertensive medication(s).
  * Cerebrovascular accident within 6 months of the first dose of study drug
* 22. Has a history of, or a current bleeding or thrombotic disorders or participants at risk for severe haemorrhage. The degree of tumour invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe haemorrhage associated with tumour shrinkage/necrosis following lenvatinib therapy.
* 23. Participants with a >1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
* 24. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* 25. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* 26. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | From baseline to 6 weeks planned resected tumour site(s) at week 6 surgery
  Proportion of patients with complete absence of residual melanoma cells in the the planned resected tumour site(s) at week 6 surgery.
The anti-tumoural immune response | Baseline, week 1 week 6
  Changes in T cell tumour infiltration, tumour PD-L1 expression, melanoma antigen expression, presence of regulatory T cells, immunosuppressive cytokines, VEGF signalling and modulation of the tumour vasculature.

SECONDARY OUTCOMES:
Objective clinical (RECIST) response rate | From baseline to 6 weeks
  Proportion of patients with complete and partial responses at 6 weeks compared to baseline per RECIST guidelines for each treatment arm.
Metabolic response rate | From baseline to 6 weeks
  Proportion of patients with complete and partial metabolic responses assessed by PET scan at 6 weeks compared to baseline for each treatment arm.
Relapse free survival | 10 years
  The amount of time that patients are disease free from the time of surgery at 6 weeks from study entry.
Treatment free survival | 1, 2, 3, 4, 5 and 10 years from the end of adjuvant treatment
  The proportion of patients who have not had a relapse of disease during study treatment and who have no requirement for new melanoma treatment from the end of adjuvant treatment period.
Overall survival | 10 years
  The proportion of patients who are alive from the time of study entry
Incidence of post operative infection | 6 weeks
  The number of patients (and the number of episodes) who develop a post operative infection of the surgical wound requiring intravenous antibiotics and/or wound drainage.
Incidence of post operative seroma formation | 6 weeks
  The number of patients (and the number of episodes) who develop a seroma at the surgical site that requires any intervention and the volume of seroma drainage.
Duration of post operative wound drainage time | 6 weeks
  The number of days that a wound drain remains in situ from the time of surgery.
Incidence of post operative bleeding requiring return to theatre or transfusion | 6 weeks
  The number of patients (and the number of episodes) who have a bleed from the post operative surgical wound that requires a blood transfusion or return to theatre to stop the bleeding.
Comparison of surgeon's opinion of operability evaluated at baseline to time of surgery | 6 weeks
  The change, if any, in the surgeon's assessment of 'operability' from baseline opinion (based on clinical and imaging examination) to time of operation.
Incidence of any treatment-emergent adverse events | 52 weeks
  The number of study treatment related adverse events of all Common Terminology Criteria for Adverse Events (CTCAE) grades from the time of starting study treatment to the time of permanent discontinuation of study treatment.
Description of the morphological assessment of melanoma tissue | Baseline, week 1, week 6
  The effects of study treatment on the degree of necrosis and genetic markers in tumour tissue prior to surgery.
Description of the RNA expression profile of melanoma tumour | Baseline, week 1, week 6
  The effects of study treatment on the baseline function of RNA expression in tumour tissue prior to surgery.
Measurement of leucocyte subpopulations in peripheral blood | Baseline, week 1, week 6
  The effects of study treatment on the number and type of white cells in the blood.
Measurement of circulating tumour DNA | Baseline, week 1, week 6
  The levels of melanoma DNA that is circulating in the blood stream and the changes during study treatment.
Concordance of metabolic response measured by pathological response | 6 weeks
  The activity of melanoma tissue assessed by the uptake of fludeoxyglucose (18F) in tumour cells viewed using positron emission tomography (PET) and how well this corresponds to the findings from the pathological examination of completely excised tumour tissue.
Concordance of metabolic response measured by RECIST response | 52 weeks
  The activity of melanoma tissue assessed by the uptake of fludeoxyglucose (18F) in tumour cells viewed using positron emission tomography (PET) and how well this corresponds to the assessment of tumour size and extent using computed tomography and magnetic resonance imaging scans.
Concordance of pathological response measured by RECIST response | 6 weeks
  The findings from the pathological examination of completely excised tumour tissue and how well this corresponds to the assessment of tumour size and extent using computed tomography and magnetic resonance imaging scans
Concordance of metabolic response with RECIST response at relapse | 52 weeks
  The activity of recurrent melanoma tissue assessed by the uptake of fludeoxyglucose (18F) in tumour cells viewed using positron emission tomography (PET) and how well this corresponds to the assessment of tumour size and extent using computed tomography and magnetic resonance imaging scans.
Quality of life scores | At baseline, weeks 6, 15, 21, 27, 33, 39, 45, 51
  The individual, summary and composite scores obtained from the validated EUROQOL QLQ-C30, EQ-5D and FACT-M questionnaires

OTHER OUTCOMES:
Concordance of immune related response criteria (irRC) with RECIST response | Weeks 6 and 52
  The application of two different criterion to establish the tumour burden as assessed with computed tomography and magnetic resonance imaging.
Correlation of the gut microbiome with RECIST response to immunotherapy | Baseline, Week 6, week 24, at relapse if this occurs within 10 years from study entry
  Characterisation of the bacterial diversity and composition in stool samples at baseline, prior to surgery at week 6, week 24 and at relapse.
Correlation of intestinal permeability with treatment response and toxicity | Baseline and during 52 weeks of treatment
  Degree of intestinal mucosal integrity measured by the ability of two non-metabolized sugar molecules (lactulose and mannitol) recovered in a urine sample collected over 6 hours following ingestion.
Characterisation of self-reported dietary habits (including use of oral probiotics) and correlation with the gut microbiome | Baseline
  Diet plays a significant role in shaping the intestinal microbiome. Nutrition may influence the gut microbiome and response to immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina V Long, Study Director — Melanoma Institute Australia
Locations (1):
- Melanoma Institute Australia, North Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No